CLINICAL TRIAL: NCT06880809
Title: Bridging the Gap: A Collaborative Intervention Group for Black Youth at Risk for Suicide
Brief Title: Bridge the Gap (BTG) - Black Youth Group
Acronym: Bridge the Gap
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Tia Tyndal, Principle Investigator, Psychology Postdoctoral Fellow, Children's Hospital Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CHLA-25-00072
Record Dates: First submitted 2025-03-12; First posted 2025-03-18 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Suicide Prevention
Keywords: Suicide Prevention; Black Youth; Collaborative Assessment & Management of Suicidality (CAMS); Group Intervention
MeSH Terms: conditions — Suicide Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Arm (Experimental): Participants will complete a 10-week group and complete pre-treatment and post-treatment assessment measures.
  Interventions: Behavioral: Bridge the Gap (BTG) - Black Youth Group

INTERVENTIONS:
Behavioral: Bridge the Gap (BTG) - Black Youth Group — Participants will complete a group intervention, rooted in the Collaborative Assessment & Management of Suicidality (CAMS) evidence-based model, driven by their own unique identification of suicide drivers.

SUMMARY:
The goal of this clinical trial is to develop and preliminarily test a culturally adapted suicide intervention specifically for black youth. The main question it aims to answer:

-To evaluate the feasibility and acceptability of the group, as well as the preliminary efficacy of the group for decreasing suicidal thoughts and behaviors and increasing protective factors such as hope, positive ethnic identity, and family and peer support.

Participants will be asked to attend 10-week group intervention and complete pre-treatment and post-treatment assessment measures.

ELIGIBILITY:
Inclusion Criteria:

* 12-17 years old
* Identify as Black or African American or being of African descent
* Have current suicidal ideation or suicidal ideation within the last 30 days
* Have assent from the adolescent participant and consent from an individual's caregiver or guardian to participate.

Exclusion Criteria:

* An active psychotic disorder or current psychosis symptoms
* No history of suicide attempt(s) or suicide ideation in the past 30 days
* Cognitive deficits or a medical condition diagnosed from a medical provider that precludes full understanding of study materials as assessed through an inability to complete the pre-treatment CAMS SSF & SSP
* Caregivers, guardians, and/or the patient refuse to participate.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 16 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The Collaborative Assessment & Management of Suicidality - Suicide Status Form (SSF) | From pre-treatment until 3 months post-treatment, approximately 23 weeks.
  An assessment of suicide risk that consists of six core assessment constructs: psychological pain, stress, agitation, hopelessness, self-hate, and overall risk of suicide; as well as reasons for living and reasons for dying constructs, and wish to live and wish to die constructs.
Ethnic Identity Scale (EIS) | From baseline until 3 months post-treatment, approximately 22 weeks.
  A 17-item scale that assesses the three components of ethnic identity and distinguishes between exploration, resolution, and affirmation. Scores range from 17-68, with higher scores indicating higher levels of affirmation, exploration, and resolution.
Living Ladder Scale | From baseline until 3 months post-treatment, approximately 22 weeks.
  A one-item measure that is prospectively associated with suicidal ideation and suicide attempts by measuring readiness to continue living among individuals thinking of suicide. Scores range from 0-8, with 8 indicating an individual is committed to making changes to make their lives worth living.
Brief Suicide Cognitions Scale (B-SCS) | From baseline until 3 months post-treatment, approximately 22 weeks.
  A 6-item self-report scale that measures the suicidal belief system, including dimensions of unlovability, unbearability, and unsolvability. Scores range from 6-30, with lower scores indicating fewer suicide cognitions.
Therapeutic Relationship Working Alliance Inventory, Short Revised (WAI-SR) | From baseline until 3 months post-treatment, approximately 22 weeks.
  A 12-item scale that reflects Bordin's three-dimensional conceptualization of therapeutic alliance: task, goal, and bond. Scores range from 12-60, with higher scores indicating higher therapeutic alliance.
Optimism and Hope Scale (OHS) | From baseline until 3 months post-treatment, approximately 22 weeks.
  A 14-item scale that measures an individual's level of both optimism, as characterized by a positive outlook on the future, and hope, as characterized by the belief in one's ability to achieve goals and navigate challenges. Scores range from 14-56, with lower scores indicating more hope and optimism.
Parent Readiness for Hospital Discharge Scale (RHDS) | From baseline until 3 months post-treatment, approximately 22 weeks.
  A 23-item scale aimed at providing a discharge readiness assessment before pediatric discharge from care in hospital settings. Scores range from 0-80, with higher scores indicating more readiness.
Group Cohesion Scale | From baseline until the beginning of post-treatment, approximately 10 weeks.
  A 12-item self-report scale that measures group cohesion, including dimensions of engagement, conflict, and avoidance. Scores across the subscales range from 0-72; higher scores indicate more of that dimension.

CONTACTS AND LOCATIONS:
Overall Officials: Tia Tyndal, PhD, Principal Investigator — Children's Hospital Los Angeles

IPD SHARING:
Plan to Share IPD: No